CLINICAL TRIAL: NCT04345029
Title: Randomized Controlled Trial of Efficacy of a Natural Ingredient on Appetite Regulation in Overweight / Obese Patients Grade I
Brief Title: Effectiveness of a Natural Ingredient on Appetite Regulation
Acronym: SAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-00012
Record Dates: First submitted 2020-04-06; First posted 2020-04-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-04

CONDITIONS: Appetite Regulation; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Lippia citriodora + sabdariffa) (Experimental): Consumption for 60 days of Lippia citriodora 325 mg + Hibiscus sabdariffa 175 mg.
  Two capsules per day will be consumed thirty minutes before breakfast orally for 60 days.
  Interventions: Dietary Supplement: Dietary supplement consumption
- control group Placebo (sucrose) (Placebo Comparator): Two capsules per day will be consumed thirty minutes before breakfast orally for 60 days.
  Interventions: Dietary Supplement: Dietary supplement consumption

INTERVENTIONS:
Dietary Supplement: Dietary supplement consumption — The experimental product consumption time was 60 days and the control consumption time was 60 days.
  Each subject must consume both products, with a washing period of 30 days.

SUMMARY:
Single-center, double-blind, double-crossed, randomized controlled clinical trial with two crossed branches, designed with the objective of evaluating the effect of the investigational product on satiety.

DETAILED DESCRIPTION:
Subjects who meet the selection criteria will make a total of five visits to the research laboratory and will carry out the tests established in the protocol. Subsequently, a statistical analysis will be performed with the variables measured in the study to obtain results.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Both genders.
* BMI 25-34.9 kg / m2, both inclusive.
* Weight maintained during the last 3 months.
* Smoking subjects or not, but in any case they do not change their nicotinic habits during their participation in the study.
* Absence of disease diagnosed at the start of the study.

Exclusion Criteria:

* Thyroid dysfunction, infections, or with any type of chronic disease (eg, autoimmune, inflammatory).
* History of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Subjects who are performing or intend to carry out any type of diet, low-calorie or not, during the study.
* Participation in another clinical trial in the three months prior to the study.
* Lack of will or inability to comply with clinical trial procedures.
* Pregnant woman.
* Subjects whose condition does not make them eligible for the study according to the researcher's criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Evolution of appetite sensation | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in eva scale (%)
Sensation of appetite before intaking the product under investigation | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in eva scale (%)
Area under the curve of the evolution of the appetite sensation from instant zero ingestion to instant ingestion of 60 minutes | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in eva scale (%)
Average of the appetite sensation during the 60 minutes after intake of the experimented product | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in eva scale (%)
Decrease in the sensation of appetite suffering from subjects when consuming the product in experimentation | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in eva scale (%)
Area under the curve of the evolution of the appetite feeling from the 60 minutes post-intake instantly 240 minutes post-intake. | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in eva scale (%)
Appetite sensation at 240 minutes post-ingestion and area under the curve of the evolution of appetite feeling from instant zero post-intake to instant 240 minutes post-intake | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in eva scale (%)
Appetite feeling immediately after ad-libitum food | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in eva scale (%)
Amount of energy consumed during the ad-libitum meal | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in kcal with the weighing of the food consumed in the ad libitum test
Satiety quotient (SQ) | It is measured twice, both at the end of taking the product after 60 days (placebo and experimental product)
  Satiety assessment, measured in kcal with the weighing of the food consumed in the ad libitum test

SECONDARY OUTCOMES:
Insulinemia | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product. And in the ad libitum test.
  Hormonal analysis, measured in mU/L
Leptin | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product. And in the ad libitum test.
  Hormonal analysis, measured in ng/dL
Adiponectin | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product. And in the ad libitum test.
  Hormonal analysis, measured in µg/mL
Ghrelin (GHRL) | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product. And in the ad libitum test.
  Hormonal analysis, measured in ng/ml
Tyrosine Peptide Tyrosine (PYY) | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product. And in the ad libitum test.
  Hormonal analysis, measured in pg/mL
Glucagon Like Peptide - 1 (GLP-1) | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product. And in the ad libitum test.
  Hormonal analysis, measured in ng/mL
Blood glucose | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product. And in the ad libitum test.
  Glycidic analysis, measured in mg/dL
Glycosylated hemoglobin (HBA1c) | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Glycidic analysis, measured in %
Peripheral insulin resistance (HOMA-IR) | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Glycidic analysis
Total Cholesterol | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Lipidic profile, measured in mg/dl
LDL - Cholesterol | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Lipidic profile, measured in mg/dl
HDL - Cholesterol | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Lipidic profile, measured in mg/dl
Triglycerides | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Lipidic profile, measured in mg/dl
Fat mass | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Bioimpedance, in Kg. For this we will use a TANITA
Muscle mass | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Bioimpedance, in Kg. For this we will use a TANITA
Body mass index | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  Bioimpedance, in Kg/m2. For this we will use a TANITA
Physical activity | It will be measured for 3 days before and after the consumption time (60 days) with the experimental product and the placebo product.
  Measured in MET, with Actigraph wGT3X-BT
Gastrointestinal Quality of Life Test | It is measured before and after the consumption time (60 days) with the experimental product and the placebo product.
  GIQLI
Quality of Life Test | It is measured before and after the consumption time (60 days) with the experimental product and the placebo product.
  WHOQOL BREF
Liver safety variables | It is measured on an empty stomach, before and after the consumption time (60 days) with the experimental product and the placebo product.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain